CLINICAL TRIAL: NCT02999425
Title: Effectiveness of Targeted Educational Intervention on Healthy Lifestyle Behaviors in Serbian Population: Make Right Choices Fro Lifelong Health
Brief Title: Effectiveness of Targeted Educational Intervention on Healthy Lifestyle Behaviors in Serbian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASA-1617
Record Dates: First submitted 2016-12-15; First posted 2016-12-21 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Education (Experimental): Educational intervention to study participants
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Educational intervention

SUMMARY:
The overall idea to be evaluated in this project is that educational activities providing top-notch knowledge on diet and physical activity may represent an additional benefit to the strategies aimed at decreasing lifestyle diseases in Serbian population of both young and mature age. The specific objectives of this project are:

1. to develop user-friendly guidelines for physical activity and nutrition for two age group cohorts (K-12 and adults) of Serbia residents;
2. to provide a brief educational intervention about nutrition and healthy lifestyles at school or work settings in each age group;
3. to determine if an educational intervention would yield an additional benefit in the acquisition of knowledge on nutrition and physical activity;
4. to promote and disseminate project results using popular media, non-professional and professional bodies and relevant events.

DETAILED DESCRIPTION:
In the first stage of the project, investigators will recruit national experts from academia and governmental bodies to develop distinctive user-friendly guidelines on nutrition and physical activity based on gold-standard recommendations currently available, from the US Centers for Disease Control and Prevention, World Health Organization, American College of Sports Medicine and American Heart Association. Intended for general public, two laymen guidelines will be produced, each for a specific age group (K-12 and adults), with both documents outline how people can improve their overall eating patterns and how children and adults can improve their health through physical activity. For the second stage, ~ 2.000 participants (a nationally representative sample of K-12 and adult age group) will participate in a tailored educational intervention delivered by CHESS experts (health professional and physical education teachers), with a summary of above layman reports delivered to recruited participants via 50 oral sessions. Both groups will complete pre- and post-intervention questionnaires of the Health-Promoting Lifestyle Profile (HPLS) and Short-Form Health Survey, standard easy-to-administer questionnaires that measure health-promoting lifestyle knowledge in different scales. In the third phase, investigators will compare the effectiveness of targeted health-promoting education, comparing pre-intervention vs. post-intervention (at 3 months) HPLS total scores. Collected data will be organized in nationally recognized Open Access database, with descriptive information on all relevant outcomes presented in user-friendly electronic format for whole sample and each age-specific sub-population. Finally, both guidelines on nutrition and physical activity, and the outcomes on educational intervention to promote healthy lifestyles among K-12 and adult population will be further disseminated:

1. to general public through media, conferences and Layman's report;
2. to interested and relevant stakeholders in the field of health, education and sport through overview in brief memorandum; and
3. to professional bodies and groups through interactive meetings and workshops.

Finally, the results will be further disseminated at relevant conferences, e-media and journal papers.

ELIGIBILITY:
Inclusion Criteria:

* General population older than 10 years

Exclusion Criteria:

* Clinical patients

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3822 (Actual)
Dates: Start 2016-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Knowledge assessed on the Health-Promoting Lifestyle Profile | Change from Baseline Knowledge at 3 months

SECONDARY OUTCOMES:
Health-Related Quality of Life assessed on the Short-Form Health Survey | Change from Baseline Health-Related Quality of Life at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sergej M Ostojic, MD, PhD, Study Chair — Center for Health, Exercise and Sport Sciences
Locations (1):
- Center for Health, Exercise and Sport Sciences, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Assessed outcomes will be shared via open database when study finished, via direct contact with PI

REFERENCES:
- [Background] Holt AM, Jancey J, Lee AH, Kerr DA, Hills AP, Anderson AS, Howat PA. A cluster-randomised controlled trial of a physical activity and nutrition programme in retirement villages: a study protocol. BMJ Open. 2014 Sep 25;4(9):e005107. doi: 10.1136/bmjopen-2014-005107. PMID 25256185
- [Background] Gillison F, Standage M, Verplanken B. A cluster randomised controlled trial of an intervention to promote healthy lifestyle habits to school leavers: study rationale, design, and methods. BMC Public Health. 2014 Mar 4;14:221. doi: 10.1186/1471-2458-14-221. PMID 24592967
- [Background] Morgan PJ, Collins CE, Plotnikoff RC, Callister R, Burrows T, Fletcher R, Okely AD, Young MD, Miller A, Lloyd AB, Cook AT, Cruickshank J, Saunders KL, Lubans DR. The 'Healthy Dads, Healthy Kids' community randomized controlled trial: a community-based healthy lifestyle program for fathers and their children. Prev Med. 2014 Apr;61:90-9. doi: 10.1016/j.ypmed.2013.12.019. Epub 2013 Dec 29. PMID 24380796